CLINICAL TRIAL: NCT02390960
Title: A Phase 2a, Single-Dose, Double-Blind, Placebo-Controlled, 2-Way Crossover Study to Evaluate the Efficacy and Safety of SST-6006 Compared to Placebo in the Treatment of Erectile Dysfunction
Brief Title: Phase 2a Topical Sildenafil Proof-of-Concept Study in Men With Mild to Moderate ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SST-6006-007-01
Record Dates: First submitted 2015-03-09; First posted 2015-03-18 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil (SST-6006) is a preserved, white to off-white, topical cream. The active ingredient is 5% sildenafil citrate by weight. During the SST-6006 dosing period, penile plethysmography will be utilized to evaluate efficacy of SST-6006 verses placebo cream. The plethysmography session will be approximately 75 minutes. This includes a 15 minute 'baseline' period where patients are told to remain in the flaccid state and 60 minutes during which time patients will watch a series of erotic videos.
  Interventions: Drug: Sildenafil Cream; Device: Penile Plethysmography (RigiScan)
- Placebo (Placebo Comparator): Placebo cream will be the same as SST-6006 without the active ingredient, sildenafil citrate. It will be matched in appearance, smell, consistency, and color to SST-6006 topical sildenafil cream. During the placebo cream dosing period, penile plethysmography will be utilized to evaluate efficacy of SST-6006 verses placebo cream. The plethysmography session will be approximately 75 minutes. This includes a 15 minute 'baseline' period where patients are told to remain in the flaccid state and 60 minutes during which time patients will watch a series of erotic videos.
  Interventions: Drug: Placebo Cream; Device: Penile Plethysmography (RigiScan)

INTERVENTIONS:
Drug: Sildenafil Cream — Patients will be instructed to apply pre-weighed SST-6006 to the non-erect penile skin area at the time of dosing. Patients will then massage the cream into the penile shaft and glans for a maximum of 3 minutes.
  Other Names: SST-6006
  Arms: Sildenafil
Drug: Placebo Cream — Patients will be instructed to apply the pre-weighed placebo cream to the non-erect penile skin area at the time of dosing. Patients will then massage the cream into the penile shaft and glans for a maximum of 3 minutes.
  Arms: Placebo
Device: Penile Plethysmography (RigiScan) — During each dosing period, penile plethysmography will be utilized to evaluate efficacy of SST-6006 verses placebo cream. Each plethysmography session will be approximately 75 minutes.This includes a 15 minute 'baseline' period where patients are told to remain in the flaccid state and 60 minutes during which time patients will watch a series of erotic videos.

SUMMARY:
This is a Phase 2a, single-dose, double-blind, placebo-controlled, 2-way crossover study in men with ED. A single 2 gram dose of SST-6006 topical cream 5% w/w (formulated to deliver 100 mg of sildenafil) or a topical placebo cream will be applied to the penile shaft and glans. There are 4 study phases: the Initial Patient Screening Phase (Visit 1, an Off Site 4-Week Run-in Period and Visit 2), the Final Patient Screening Phase (Visit 3), the SST-6006/Placebo Double-Blind Dosing Phase (Visits 4-5), and the Follow-up Phase. Primary outcomes will be be evaluated at Weeks 7 and 8 of the study

DETAILED DESCRIPTION:
Initial Patient Eligibility: Visit 1 (Day 1) After the patient provides written informed consent, the initial screening procedures will be performed. Patients who meet all eligibility criteria will be instructed on completion of the SEP Diary, the need for a one week washout of any ED medications before starting the Off-Site 4-Week Run-In Period and that the use of any ED medications will be prohibited throughout the entire 4-week duration and up until the completion of Visit 5. Site staff will contact patients by phone between 4 and 7 days following Visit 1 (on Days 4- 7) to communicate eligibility (met laboratory parameters and the one week washout) to participate in the Off-Site 4-Week Run-In Period. Site staff will also schedule the Topical Placebo RigiScan Qualification Visit (Visit 2) to be within two days of completion of the 4-Week Run-In Period for eligible patients. Ineligible patients will be instructed to discard their SEP Diary and will be discontinued from further study participation Off-Site 4-Week Run-In Period (Day 8-35) Eligible patients will participate in an Off-Site 4-Week Run-In Period during which time they will attempt intercourse a minimum of 4 times. Use of any ED medications will be prohibited throughout the entire 4-week duration and up until the completion of Visit 5. Patients will be asked to maintain a Sexual Encounter Profile (SEP) diary during the 4-Week Run-In Period to be completed after each intercourse attempt.

Topical Placebo RigiScan Qualification: Visit 2 (Day 36 [+ 2 days]) Patients who successfully complete the 4-Week Run-In will be instructed to complete the IIEF questionnaire at the beginning of Visit 2. Eligible patients must have documented mild-moderate ED as demonstrated by a score of 11-21 in the International Index of Erectile Function (IIEF) Erectile Function domain of the IIEF questionnaire.

Eligible patients will then complete a single-blind (patient) 60 minute plethysmography procedure using placebo cream to familiarize patients with the plethysmography device (i.e. RigiScan) and evaluate the placebo response with Visual Sexual Stimulation (VSS).

Patients who demonstrate a topical placebo response (i.e. achieve an erection of ≥ 60% rigidity at the base of the penis for a cumulative duration of > 4 minutes) will be ineligible for further study participation. Any patients with an adverse dermatologic reaction to the placebo cream will be excluded from further participation in the study but will be followed until normalization of symptoms.

Safety data for all patients, regardless of continued eligibility, will be included in the database as patients will have been exposed to IP (placebo cream only) during this visit. There will be a 7 (± 1) day washout period between Visits 2 and 3.

Oral Sildenafil RigiScan Qualification: Visit 3 (Day 43 [± 2 days]) Patients who meet the eligibility criteria will then complete the Oral Sildenafil RigiScan Qualification visit, consisting of a single-blind (patient) plethysmography procedure with 60 minutes of VSS to evaluate the patient's response to oral sildenafil.

Patients who do not respond to oral sildenafil (i.e., do not achieve ≥ 60% rigidity at the base of the penis for a cumulative duration of >15 minutes and an EHS Score of 3 or 4) will be excluded from further study participation.

There will be a 7 (± 1) day washout period between Visit 3 and Visit 4 (i.e., the first visit in the SST-6006/Placebo Double-Blind Dosing Phase).

SST-6006/Placebo Double-Blind Dosing Phase: Visits 4 & 5 (Days 50 and 57 [± 2 days]) Eligible patients will be randomized to a sequence of dosing (i.e., placebo cream then SST-6006 or SST-6006 then placebo cream). The SST-6006/Placebo Double-Blind Dosing Phase will consist of two plethysmography procedures with 60 minutes of VSS. One will evaluate the patient's response to SST-6006 and the other will evaluate the patient's response to placebo cream. Patients will be instructed to complete a 4-Point Erection Hardness Scale (EHS) immediately following completion of the plethysmography procedure at each visit. There will be a 7 (± 1) day wash-out between Visit 4 and Visit 5.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a heterosexual male ≥ 18 and ≤ 70 years of age.
2. Patient has had a clinical diagnosis of erectile dysfunction for a minimum of 6 months.
3. Patient has a body mass index (BMI) from 18 to 30 kg/m², inclusive.

5. Patient is capable of understanding and complying with the protocol and agrees to sign the informed consent document.

6 Patient agrees to use condoms with sexual activity for 7 days immediately following each visit that involves application of SST-6006 or placebo cream (i.e. Visit 2, Visit 4 and Visit 5).

7. Patient has a testosterone level ≥ 300 ng/dL (either naturally or through androgen replacement therapy; if on androgen replacement therapy, must have been taking for ≥ 6 months).

8. Patient is willing to undergo plethysmography procedure with VSS during the trial

-

Exclusion Criteria:

Subject is unfamiliar with or unwilling to watch visual sexual stimulation (VSS).

2. Subject has any disorder or a history of any disorder that may prevent the successful completion of the study.

3. Subjects with an abnormal physical exam, that in the opinion of the Investigator, would interfere with study participation.

4. Subject has a significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or psychiatric disease or other unstable medical condition that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, contraindicate sexual activity, or confound the interpretation of study results.

5. Subject has an active ulcer or clinically significant bleeding disorder. 6. Subject has a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to Visit 1; a history of coronary disease causing angina; or congestive heart failure requiring medical intervention.

7. Subject has uncontrolled hypertension or untreated hypertension. 8. Subject has a history of orthostatic hypotension or orthostatic hypotension.

9. Subject is unable to walk up and down two flights of stairs briskly without chest pain.

10. Subject is using alpha blockers. 11. Subject is using or has possession of nitrate containing medication(s). 12. Subject has retinitis pigmentosa or sickle cell anemia or related anemias, even if the subject feels clinically well at the time of screening. Subjects with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning subjects as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history.

13. Subject has anatomical deformation of the penis such as angulation, cavernosal fibrosis, or Peyronie¡-s disease, or history of genital surgery.

14. Subject has a history of prostate surgery. 15. Subject has a history of pelvic radiation. 16. Subject has type 1 or type 2 diabetes. 17. Subject has a history of cancer other than basal cell carcinoma. 18. Subject has any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article.

19. Subject has a history of drug abuse within 1 year before Visit 1. 20. Subject has a history of alcoholism within 1 year before Visit 1, admitted alcohol abuse, or has an average consumption of more than 2 standard units of alcohol per day (a standard unit equals 12 ounces of beer, 1¨ö ounces of 80-proof alcohol, or 6 ounces of wine).

21. Subject has had treatment currently or within 1 month (28 days) of Visit 1 with any of the following: weak, moderate, and strong inhibitors and inducers of CYP3A4 and CYP2C9 enzymes (e.g., CYP3A4: ketoconazole, clarithromycin, verapamil, diltiazem, St. John¡-s Wort / CYP2C9: fluconazole, oxandrolone, fluvastatin, and metronidazole). Any prescription, over-the-counter (OTC) medications, or herbal products taken recently or currently being taken will be screened by study personnel prior to study enrollment to confirm such drugs do not inhibit or induce the two enzymes listed above. If the subject takes any prescription or OTC drugs at the direction of a health care provider that are inhibitors or inducers of CYP3A4 and CYP2C9, that provider should be consulted before medications are stopped for the purposes of study participation.

22. Subject is unwilling to refrain from using any medication for erectile dysfunction, with the exception of study medication, after Visit 1 and throughout the duration of the study up until the completion of Visit 5.

23. Subject has positive findings from urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, and opiates).

24. Subjects with a positive alcohol breath test. 25. Subject participated in any clinical research study evaluating another investigational drug or therapy within 30 days before the Visit 1.

26. Subject is unwilling to refrain from ingesting grapefruit, grapefruit-containing products, Seville oranges, or products containing Seville oranges (e.g., orange marmalade) three days prior to each dosing visit.

27. Subject has any skin breaks, irritation, dermatoses, or lesions in the penile area to which the study cream will be applied.

28. Subject has a known hypersensitivity or allergy to any of the ingredients in the IP.

29. Subject has a significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or other unstable medical condition indicated by the laboratory results that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, contraindicate sexual activity, or confound the interpretation of study results.

30. Subjects who have abnormal laboratory parameters that, in the opinion of the Investigator, could confound interpretation of the study results.

31. Subjects who have positive serology findings for a sexually transmitted infection (i.e. syphilis, gonorrhea, chlamydia, HIV antibodies, hepatitis b surface antigen (HBsAg) or hepatitis c (HCV) antibodies.

32. Subjects with abnormal vital signs and/or ECG results that, in the opinion of the Investigator, would affect the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of ≥ 60% rigidity at the base of the penis during 60 minutes of VSS (SST-6006 compared to placebo cream) | 60 minutes

SECONDARY OUTCOMES:
Percentage of patients reporting occurrence of at least one Grade 3 or Grade 4 erection as defined by the EHS (refer to Appendix B) (SST-6006 compared to placebo cream) | 60 minutes
Adverse Events | From first application of cream (Week 5) through follow-up phone call (Week 9)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fossel, PhD, Study Director — Sponsor GmbH
Locations (3):
- United States (3):
  - San Diego Sexual Medicine, San Diego, California
  - Tulane Medical Center, New Orleans, Louisiana
  - Manhattan Medical Research, New York, New York